CLINICAL TRIAL: NCT01423890
Title: A Prospective Cohort Study to Evaluate the Oncotype DX® Test in Early Stage Breast Cancer
Acronym: ONCOTYPEDX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OCOG-2011-ONCOTYPEDX
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Oncotype DX; Adjuvant! Online; Decisional Conflict Scale
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Early Stage Breast Cancer (Other): Women and men with node negative, ER positive breast cancer who are receiving (or will receive) endocrine therapy, and who are candidates for chemotherapy.
  Interventions: Genetic: ONCOTYPEDX Test

INTERVENTIONS:
Genetic: ONCOTYPEDX Test — Gene signature test containing 21 genes (16 cancer-related genes, e.g., invasion, proliferation, ER, Her 2 and five reference genes) and generates an individualized recurrence score.

SUMMARY:
A prospective population-based cohort study is being conducted in Ontario to evaluate whether the performance of Oncotype DX® changes the treatment recommended and the treatment received in women or men with node negative, ER positive breast cancer who are receiving (or will receive) endocrine therapy and who are candidates for chemotherapy. One thousand eligible consenting women and men will have their tumor tissue specimen sent to Genomic Health where the Oncotype DX® assay will be performed.

DETAILED DESCRIPTION:
The evidence supporting the adoption of Oncotype DX® is relatively weak by the criteria used by the Ontario Health Technology Advisory Committee (OHTAC). There is only one small published prospective study that reports on Oncotype DX® changing clinical management. The economic models that estimated the potential advantages of using an Oncotype DX® guided treatment strategy may have overestimated the benefits because they assumed that all patients with tumors >1cm in the absence of Oncotype DX® testing would receive chemotherapy in addition to tamoxifen, and that the magnitude of benefit with chemotherapy over tamoxifen is relatively large, i.e. reduces recurrence risk by 74% and associated with an absolute benefit of 28%. (The benefit comes from one trial and is applied to all patients). It is estimated that there are about 3,300 incident cases with node negative, ER positive, HER2 neu negative tumors annually in Ontario, it is important to evaluate the adoption of this test for decision making in Ontario.

ELIGIBILITY:
Inclusion Criteria:

* Women or men with histologic evidence of invasive breast cancer (ductal, lobular or mixed disease).
* Surgical resection including breast conserving surgery or modified radical mastectomy or simple mastectomy, within the last four months.
* Axillary lymph nodes assessed for tumor by:

  (i) sentinel node biopsy, or (ii) axillary node dissection, or (iii) both
* Axillary lymph node assessment negative for cancer, or positive only for micrometastases (i.e., cancer <2mm by H&E stain).
* Tumor is estrogen receptor (ER) positive.
* Receiving or to receive adjuvant endocrine therapy (i.e., tamoxifen or aromatase inhibitor).
* Being considered for adjuvant chemotherapy.

Exclusion Criteria:

* Axillary lymph node positive for cancer.
* Patients with inoperable locally advanced breast cancer.
* Metastatic breast cancer, including local ipsilateral recurrence.
* HER2 neu positive.
* Physician/Patient unwilling to comply with study protocol.
* Inability to provide informed consent (e.g. dementia or severe cognitive impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1011 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in treatment recommendation | One month
  The primary outcome is the change in treatment recommendation by the oncologist and the change in treatment preference of the patient.

SECONDARY OUTCOMES:
Association between Oncotype DX® RS with other estimated risk calculations | One month
  The level of association between the Oncotype DX® RS with estimated recurrence risk calculated by Adjuvant! Online, as well as with traditional factors including tumor size, grade, and HER2 neu.
Change in patient decisional conflict | One month
  The change in the level of patient decisional conflict measured by the Decisional Conflict Scale (DCS). Additionally, the DCS has three subscales: uncertainty, effective decision making, and factors contributing to uncertainty. The change in each of these subscales will also be measured.
Robustness of economic model of sequential Adjuvant! Online followed by Oncotype DX®. | 6 months
  To determine the robustness of the economic model of sequential Adjuvant! Online followed by Oncotype DX®.

CONTACTS AND LOCATIONS:
Overall Officials: Mark N. Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG)
Locations (35):
- Canada (35):
  - Simcoe Muskoka Cancer Program - Royal Victoria Hospital, Barrie, Ontario
  - Quinte Healthcare Corporation, Belleville, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Brantford General Hospital, Brantford, Ontario
  - Joseph Brant Hospital, Burlington, Ontario
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Northeast Cancer Centre of Health Sciences North - Horizon Sante-Nord, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - The Credit Valley Hospital, Mississauga, Ontario
  - Stronach Regional Cancer Centre, Newmarket, Ontario
  - R.S. McLaughlin Durham Regional Cancer Centre - Lakeridge Health, Oshawa, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Grey Bruce Health Services, Owen Sound, Ontario
  - Peterborough Regional Health Centre, Peterborough, Ontario
  - Mackenzie Health, Richmond Hill, Ontario
  - Bluewater Health, Sarnia, Ontario
  - Algoma District Cancer Program - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Rouge Valley Health System, Scarborough Village, Ontario
  - The Scarborough Hospital, Scarborough Village, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - North York General Hospital, Toronto, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - St. Joseph's Healthcare, Toronto, Ontario
  - Trillium Health Centre, Toronto, Ontario
  - Humber River Regional Cancer Centre, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario